CLINICAL TRIAL: NCT03348163
Title: Bictegravir, Emtricitabine and Tenofovir Alafenamide in Transwomen for Optimization of ART: The (mo)BETTA Trial
Brief Title: (mo)BETTA Trial in Transwomen for Optimization of ART
Acronym: (mo)BETTA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of ability to recruit due to COVID-19 pandemic
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Jordan Elizabeth Lake, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-17-0480
Record Dates: First submitted 2017-11-08; First posted 2017-11-20 (Actual); Results first posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: HIV Infections
Keywords: Transgender women; Bictegravir
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Switch ART (Experimental): Switch from current antiretroviral therapy (ART) to bictegravir + tenofovir alafenamide + emtricitabine (B/FTC/TAF) for 48 weeks
  Interventions: Drug: B/FTC/TAF
- Continue Current ART (Active Comparator): Continue current antiretroviral therapy (ART) therapy (which is emtricitabine plus tenofovir disoproxil fumarate or tenofovir alafenamide plus 3rd agent) for 48 weeks.
  Interventions: Drug: Current ART

INTERVENTIONS:
Drug: B/FTC/TAF — B/FTC/TAF is bictegravir + tenofovir alafenamide + emtricitabine in one pill (single tablet regimen)
  Arms: Switch ART
Drug: Current ART — Current ART is emtricitabine plus tenofovir disoproxil fumarate or tenofovir alafenamide plus 3rd agent.
  Arms: Continue Current ART

SUMMARY:
The purpose of this study is to determine the safety and tolerability of a new HIV medication, bictegravir plus emtricitabine plus tenofovir alafenamide (B/FTC/TAF, 3 HIV medications combined into one pill) in HIV-infected transgender women (TW).

ELIGIBILITY:
Inclusion Criteria:

* Self-identified transgender woman (TW)
* HIV infection
* Undetectable HIV viral load (HIV-1 RNA <50 copies/mL) at screening and for >/=24 weeks prior to entry.
* Current HIV treatment with FTC plus TDF or TAF and a 3rd agent.
* No changes in ART in the 12 weeks prior to screening.
* Current female hormone therapy use.
* Ability and willingness of subject to provide informed consent.

Exclusion Criteria:

* Current or planned use of prohibited medications (Phenobarbital, Phenytoin, Carbamazepine, Oxcarbazepine, Rifampin, Rifapentine, St. John's Wort, Echinacea, Dofetilide, Cisapride, Atazanavir)
* Change or initiation of lipid- and/or glucose-lowering therapy in the 12 weeks prior to entry, or planned need for such therapy during the study period.
* Current use of androgen therapy.
* Intent to significantly modify diet or exercise habits, or to enroll in a weight loss intervention during the study period.
* Anticipated need to initiate or change doses of medications with anti-inflammatory properties within the study period.
* Screening laboratory values as follows: (ANC <500 cells/mm^3; Hemoglobin <10 gm/dL; Cr Cl <30 mL/min (estimated by CKD-Epi equation); AST or ALT >3x ULN)
* Evidence of resistance to any component of the current ART regimen (genotypic or phenotypic)
* Current use of bictegravir in another investigational setting
* Current use of other investigational agents that the participant could not receive unchanged, if needed, throughout the study period (unless approved by the study team)
* Any condition that the study investigator believes would make the candidate unsuitable for participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified transgender women (TW)
Enrollment: 26 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan E Lake, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Thomas Street Health Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 26 enrolled participants, 21 met inclusion criteria and were randomized.
Groups:
- Switch ART: Switch from current antiretroviral therapy (ART) to B/FTC/TAF for 48 weeks
  B/FTC/TAF: B/FTC/TAF in one pill (single tablet regimen) for administration to participants in Arm A.
- Continue Current ART: Continue current (ART) therapy (emtricitabine plus tenofovir disoproxil fumarate or tenofovir alafenamide plus 3rd agent) for 48 weeks
  Current ART: Comparator arm. Participant continues open label entry ART.
Period: Overall Study
Arm/Group | Switch ART | Continue Current ART
Started | 12 | 9
Completed | 10 | 9
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Switch ART | Continue Current ART | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10) | 47 (3) | 45.85 (7.85)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Self-identified transgender women (TW) | 12 | 9 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 9 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latina | 7 | 4 | 11
  White | 0 | 1 | 1
  Black/African American | 3 | 2 | 5
  Asian | 2 | 0 | 2
  Alaskan Native/American Indian | 0 | 2 | 2
  Native Hawaiian/ Pacific/Islander | 0 | 0 | 0
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Maintaining Undetectable HIV-1 RNA
Description: Number of participants who maintain <50 copies/mL HIV-1 RNA for 48 weeks
Time Frame: 48 weeks
Population: Per the protocol, participants who have to discontinue study drug early but have been on study drug for at least 12 weeks will undergo a final evaluation at the time they discontinue. One participant in the Switch ART arm discontinued the study early at 36 weeks, and data was collected for this participant at 36 weeks--this 36-week data is included in the analysis of the 48 week timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
Participants | 10 | 8

2. Primary Outcome: Frequency of Adverse Events
Description: Number of participants who discontinue study drug due to study-drug related adverse events (AEs, includes >/= Grade 3 lab or clinical events)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
Participants | 0 | 0

3. Secondary Outcome: Fat Mass, Total
Description: Fat mass, total, as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: pounds (lbs)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
pounds (lbs) | 53.49 [49.16 to 59.08] | 55.41 [52.83 to 72.79]

4. Secondary Outcome: Fat Mass, Total
Description: Fat mass, total, as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pounds (lbs)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
pounds (lbs) | 62.07 [53.12 to 71.29] | 71.57 [47.22 to 77.42]

5. Secondary Outcome: Fat Mass, Trunk
Description: Fat mass, trunk, as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: pounds (lbs)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
pounds (lbs) | 30.80 [27.82 to 38.14] | 42.21 [22.34 to 46.90]

6. Secondary Outcome: Fat Mass, Trunk
Description: Fat mass, trunk, as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pounds (lbs)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
pounds (lbs) | 34.77 [31.40 to 44.02] | 44.81 [28.99 to 53.84]

7. Secondary Outcome: Fat Mass, Limbs
Description: Fat mass, limbs, as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: baseline
Measure: Median (Inter-Quartile Range); unit: pounds (lbs)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
pounds (lbs) | 21.09 [16.19 to 23.50] | 19.60 [12.30 to 20.77]

8. Secondary Outcome: Fat Mass, Limbs
Description: Fat mass, limbs, as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pounds (lbs)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
pounds (lbs) | 23.59 [17.92 to 25.48] | 22.50 [16.33 to 35.39]

9. Secondary Outcome: Percentage of Fat Mass (Total)
Description: Percentage of Fat mass (total) as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: percentage of fat mass
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
percentage of fat mass | 33.70 [31.47 to 36.80] | 32.00 [30.80 to 38.20]

10. Secondary Outcome: Percentage of Fat Mass (Total)
Description: Percentage of Fat mass (total) as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of fat mass
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
percentage of fat mass | 35.70 [33.00 to 40.00] | 34.00 [29.60 to 44.10]

11. Secondary Outcome: Percentage of Fat Mass (Trunk)
Description: Percentage of Fat mass (trunk) as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: percentage of fat mass
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
percentage of fat mass | 40.15 [34.20 to 42.25] | 38.20 [30.35 to 41.70]

12. Secondary Outcome: Percentage of Fat Mass (Trunk)
Description: Percentage of Fat mass (trunk) as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of fat mass
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
percentage of fat mass | 41.90 [37.70 to 44.15] | 43.30 [31.20 to 45.90]

13. Secondary Outcome: Percentage of Fat Mass (Limbs)
Description: Percentage of Fat mass (limbs) as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: percentage of fat mass
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
percentage of fat mass | 57.80 [49.30 to 61.88] | 47.80 [39.85 to 58.55]

14. Secondary Outcome: Percentage of Fat Mass (Limbs)
Description: Percentage of Fat mass (limbs) as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of fat mass
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
percentage of fat mass | 59.50 [56.85 to 65.35] | 62.60 [47.20 to 71.70]

15. Secondary Outcome: Lean Mass (Total)
Description: lean mass (total) as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: pounds (lbs)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
pounds (lbs) | 108.74 [99.65 to 121.56] | 124.38 [112.11 to 146.06]

16. Secondary Outcome: Lean Mass (Limb)
Description: lean mass (limb) as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: pounds (lbs)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
pounds (lbs) | 49.79 [43.43 to 54.23] | 50.14 [47.28 to 59.86]

17. Secondary Outcome: Lean Mass (Total)
Description: lean mass (total) as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pounds (lbs)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
pounds (lbs) | 110.20 [101.34 to 116.69] | 137.37 [111.40 to 150.36]

18. Secondary Outcome: Lean Mass (Limb)
Description: lean mass (limb) as measured by Dual-energy X-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pounds (lbs)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
pounds (lbs) | 48.59 [43.53 to 55.10] | 56.34 [47.7 to 66.7]

19. Secondary Outcome: Hepatic Fat Content
Description: The controlled attenuation parameter (CAP) indicates quantity of fat in the liver (that is, hepatic fat content). CAP is assessed by performing transient elastography (TE) using a FibroScan device, which uses ultrasound. The CAP score is measured in decibels per meter (dB/m). CAP score ranges from 100 dB/m to 400 dB/m, and a higher score indicates greater hepatic fat content.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: decibel per meter (dB/m)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
decibel per meter (dB/m) | 254 [234.5 to 297.5] | 301 [271 to 318]

20. Secondary Outcome: Hepatic Fat Content
Description: as for outcome 19
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: decibel per meter (dB/m)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
decibel per meter (dB/m) | 253 [236.5 to 309.5] | 256 [235 to 294]

21. Secondary Outcome: Total Cholesterol
Description: Total cholesterol level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
milligrams per deciliter (mg/dL) | 173 [168 to 191] | 162 [148 to 180]

22. Secondary Outcome: Total Cholesterol
Description: Total cholesterol level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
milligrams per deciliter (mg/dL) | 167 [158 to 185] | 162 [156 to 171]

23. Secondary Outcome: High-density Lipoprotein (HDL) Cholesterol Level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
milligrams per deciliter (mg/dL) | 42 [38 to 50] | 44 [37 to 58]

24. Secondary Outcome: High-density Lipoprotein (HDL) Cholesterol Level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
milligrams per deciliter (mg/dL) | 54 [45 to 59] | 45 [39 to 52]

25. Secondary Outcome: Triglycerides
Description: Triglyceride level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
milligrams per deciliter (mg/dL) | 167 [96 to 335] | 90 [87 to 131]

26. Secondary Outcome: Triglycerides
Description: Triglyceride level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
milligrams per deciliter (mg/dL) | 112 [93 to 129] | 81 [74 to 145]

27. Secondary Outcome: Low-density Lipoprotein (LDL) Cholesterol Level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
milligrams per deciliter (mg/dL) | 98 [91 to 112] | 93 [79 to 104]

28. Secondary Outcome: Low-density Lipoprotein (LDL) Cholesterol Level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
milligrams per deciliter (mg/dL) | 96 [81 to 118] | 92 [92 to 95]

29. Secondary Outcome: Fasting Glucose Level
Description: Fasting Glucose level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
milligrams per deciliter (mg/dL) | 90 [86 to 99] | 92 [87 to 100]

30. Secondary Outcome: Fasting Glucose Level
Description: Fasting Glucose level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
milligrams per deciliter (mg/dL) | 86 [83 to 91] | 95 [87 to 108]

31. Secondary Outcome: Insulin Resistance
Description: The Homeostatic Assessment Model of Insulin Resistance (HOMA-IR) is an index used to determine if insulin resistance is present. HOMA-IR is calculated as ([(fasting insulin in mU/L) x (glucose in mmol/L)]/22.5). Higher HOMA-IR values indicate greater insulin resistance. The threshold HOMA-IR value that indicates insulin resistance differs among different populations, but a common clinical cutoff is 2.6 (in other words, a HOMA-IR value of 2.6 or above is commonly interpreted to indicate insulin resistance).
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: index
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
index | 2.6 [1.8 to 3.6] | 3.5 [1.3 to 9.9]

32. Secondary Outcome: Insulin Resistance
Description: as for outcome 31
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: index
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
index | 1.8 [1.1 to 3.1] | 3.9 [2 to 7.5]

33. Secondary Outcome: Oxidized Low-density Lipoprotein (LDL) Level
Description: Oxidized Low-density Lipoprotein (LDL) levels are assessed by testing blood
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Units per milliliter (U/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
Units per milliliter (U/mL) | 39859.07 [27316.60 to 53677.53] | 46282.62 [29348.98 to 51762.23]

34. Secondary Outcome: Oxidized Low-density Lipoprotein (LDL) Level
Description: Oxidized Low-density Lipoprotein (LDL) levels are assessed by testing blood
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units per milliliter
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
units per milliliter | 44375.63 [27151.89 to 46665.40] | 35476.24 [31894.04 to 45307.38]

35. Secondary Outcome: Hepatic Fibrosis as Indicated by Liver Stiffness Measurement
Description: Fibrosis (that is, scarring of the liver) results in liver stiffness, and liver stiffness can be measured by liver elastography using a FibroScan device, which uses ultrasound. The liver stiffness measurement ranges from 2 kPa to 75 kPa, with a higher score indicating greater liver scarring and stiffness
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: kilopascal (kPa)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
kilopascal (kPa) | 4.35 [4.15 to 4.45] | 4.40 [4.10 to 4.60]

36. Secondary Outcome: Hepatic Fibrosis as Indicated by Liver Stiffness Measurement
Description: as for outcome 35
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: kilopascal (kPa)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
kilopascal (kPa) | 4.30 [3.80 to 5.15] | 3.90 [3.80 to 5.10]

37. Secondary Outcome: Aspartate Aminotransferase (AST) Level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: international units per liter (IU/L)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
international units per liter (IU/L) | 20.50 [17.75 to 24.75] | 19.00 [13.00 to 26.00]

38. Secondary Outcome: Aspartate Aminotransferase (AST) Level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: international units per liter (IU/L)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
international units per liter (IU/L) | 19.00 [14.50 to 23.00] | 20.00 [14.00 to 23.00]

39. Secondary Outcome: Alanine Transaminase (ALT) Level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: international units per liter (IU/L)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
international units per liter (IU/L) | 18.50 [15.00 to 22.25] | 18.00 [14.00 to 28.00]

40. Secondary Outcome: Alanine Transaminase (ALT) Level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: international units per liter (IU/L)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
international units per liter (IU/L) | 17.00 [11.00 to 21.00] | 16.00 [13.00 to 29.00]

41. Secondary Outcome: Estimated Glomerular Filtration Rate (CKD- Epi Equations)
Description: glomerular filtration rate (GFR) level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73m^2
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
mL/min/1.73m^2 | 110.65 [97.08 to 121.93] | 105.00 [95.10 to 114.30]

42. Secondary Outcome: Estimated Glomerular Filtration Rate (CKD- Epi Equations)
Description: glomerular filtration rate (GFR) level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73m^2
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
mL/min/1.73m^2 | 102.00 [96.50 to 115.50] | 118.00 [99.00 to 119.00]

43. Secondary Outcome: Level of Adiponectin
Description: Inflammatory and metabolic biomarkers level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: nanograms per milliliter (ng/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
nanograms per milliliter (ng/mL) | 5615.81 [2760.69 to 6252.59] | 3472.11 [2444.49 to 3792.06]

44. Secondary Outcome: Level of Adiponectin
Description: Inflammatory and metabolic biomarkers level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nanograms per milliliter (ng/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
nanograms per milliliter (ng/mL) | 3120.11 [2761.61 to 5490.66] | 3681.10 [2154.24 to 5908.11]

45. Secondary Outcome: Level of Endothelin-1
Description: Inflammatory and metabolic biomarkers level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
picograms per milliliter (pg/mL) | 1.31 [1.31 to 3.73] | 3.25 [1.45 to 4.45]

46. Secondary Outcome: Level of Endothelin-1
Description: Inflammatory and metabolic biomarkers level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
picograms per milliliter (pg/mL) | 2.56 [1.73 to 3.93] | 5.23 [2.50 to 7.96]

47. Secondary Outcome: Level of Extracellular Newly Identified Receptor for Advanced Glycation End-products Binding Protein (EN-RAGE)
Description: Inflammatory and metabolic biomarkers level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
picograms per milliliter (pg/mL) | 136583.77 [83296.05 to 292690.10] | 103808.57 [77597.37 to 211495.73]

48. Secondary Outcome: Level of Extracellular Newly Identified Receptor for Advanced Glycation End-products Binding Protein (EN-RAGE)
Description: Inflammatory and metabolic biomarkers level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
picograms per milliliter (pg/mL) | 123321.76 [75937.50 to 211888.30] | 151499.70 [73791.40 to 207590.26]

49. Secondary Outcome: Level of Tumor Necrosis Factor Receptor I (TNFRI)
Description: Inflammatory and metabolic biomarkers level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
picograms per milliliter (pg/mL) | 1032.56 [957.03 to 1282.22] | 1266.15 [997.25 to 1419.70]

50. Secondary Outcome: Level of Tumor Necrosis Factor Receptor I (TNFRI)
Description: Inflammatory and metabolic biomarkers level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
picograms per milliliter (pg/mL) | 1077.17 [971.03 to 1166.63] | 1118.69 [1044.94 to 1222.00]

51. Secondary Outcome: Level of Tumor Necrosis Factor Receptor II (TNFRII)
Description: Inflammatory and metabolic biomarkers level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
picograms per milliliter (pg/mL) | 2552.35 [2042.89 to 2723.74] | 2717.57 [2235.73 to 3487.42]

52. Secondary Outcome: Level of Tumor Necrosis Factor Receptor II (TNFRII)
Description: Inflammatory and metabolic biomarkers level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
picograms per milliliter (pg/mL) | 2306.88 [2010.94 to 2930.54] | 2388.98 [2166.38 to 2541.04]

53. Secondary Outcome: Level of Insulin
Description: Inflammatory and metabolic biomarkers level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: picomoles per liter (pmol/L)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
picomoles per liter (pmol/L) | 77.08 [47.32 to 92.00] | 107.44 [35.15 to 214.51]

54. Secondary Outcome: Level of Insulin
Description: Inflammatory and metabolic biomarkers level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: picomoles per liter (pmol/L)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
picomoles per liter (pmol/L) | 52.51 [37.15 to 101.53] | 105.42 [47.75 to 193.38]

55. Secondary Outcome: Level of D-dimer
Description: Inflammatory and metabolic biomarkers level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: nanograms per milliliter (ng/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
nanograms per milliliter (ng/mL) | 193.76 [178.96 to 286.62] | 195.64 [136.32 to 264.94]

56. Secondary Outcome: Level of D-dimer
Description: Inflammatory and metabolic biomarkers level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nanograms per milliliter (ng/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
nanograms per milliliter (ng/mL) | 278.59 [198.10 to 325.27] | 197.94 [136.29 to 426.50]

57. Secondary Outcome: Level of Tissue Factor
Description: Inflammatory and metabolic biomarkers level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
picograms per milliliter (pg/mL) | 38.16 [13.39 to 72.02] | 57.73 [34.00 to 90.90]

58. Secondary Outcome: Level of Tissue Factor
Description: Inflammatory and metabolic biomarkers level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
picograms per milliliter (pg/mL) | 37.33 [12.84 to 63.28] | 44.34 [40.47 to 70.70]

59. Secondary Outcome: Level of Soluble CD14 (sCD14)
Description: Inflammatory and metabolic biomarkers level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Nanograms per milliliter
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
Nanograms per milliliter | 1369.58 [1189.94 to 1397.92] | 1447.20 [1275.56 to 1778.98]

60. Secondary Outcome: Level of Soluble CD14 (sCD14)
Description: Inflammatory and metabolic biomarkers level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Nanograms per milliliter
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
Nanograms per milliliter | 1303.36 [1177.44 to 1353.81] | 1324.06 [1132.88 to 1769.81]

61. Secondary Outcome: Level of Plasminogen Activator Inhibitor (PAI-1)
Description: Inflammatory and metabolic biomarkers level
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
picograms per milliliter (pg/mL) | 154698.40 [135732.18 to 279220.47] | 256300.04 [196833.97 to 337843.62]

62. Secondary Outcome: Level of Plasminogen Activator Inhibitor (PAI-1)
Description: Inflammatory and metabolic biomarkers level
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
picograms per milliliter (pg/mL) | 245468.27 [190452.39 to 345932.02] | 155299.95 [143319.87 to 290646.04]

63. Secondary Outcome: Bone Mineral Density (BMD), Femur Total Mean
Description: BMD as measured by dual-energy x-ray absorptiometry (DXA)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: grams per square centimeter
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
grams per square centimeter | 1.07 [0.97 to 1.10] | 0.98 [0.93 to 1.15]

64. Secondary Outcome: Bone Mineral Density (BMD), Femur Total Mean
Description: BMD as measured by dual-energy x-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: grams per square centimeter
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
grams per square centimeter | 1.07 [0.99 to 1.12] | 1.03 [0.94 to 1.17]

65. Secondary Outcome: Bone Mineral Density (BMD), AP-spine L1-L4
Description: BMD as measured by dual-energy x-ray absorptiometry (DXA)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: grams per square centimeter
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
grams per square centimeter | 1.17 [1.10 to 1.27] | 1.21 [1.16 to 1.29]

66. Secondary Outcome: Bone Mineral Density (BMD), AP-spine L1-L4
Description: BMD as measured by dual-energy x-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: grams per square centimeter
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
grams per square centimeter | 1.18 [1.09 to 1.27] | 1.24 [1.20 to 1.33]

67. Secondary Outcome: T-Score AP-spine L1-L4
Description: Bone Mineral Density T-score as measured by dual-energy x-ray absorptiometry (DXA)
  A T-score between +1 and -1 is considered normal or healthy. A T-score between -1 and -2.5 indicates osteopenia. A T-score of -2.5 or lower indicates osteoporosis
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
score on a scale | -0.20 [-1.00 to 0.40] | -0.10 [-0.50 to 0.62]

68. Secondary Outcome: T-Score AP-spine L1-L4
Description: as for outcome 67
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
score on a scale | -0.30 [-1.05 to 0.25] | 0.15 [-0.20 to 0.90]

69. Secondary Outcome: T-Score Total Body
Description: as for outcome 67
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
score on a scale | 0.05 [-0.52 to 0.55] | 0.00 [-1.00 to 1.80]

70. Secondary Outcome: T-Score Total Body
Description: as for outcome 67
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
score on a scale | -0.10 [-0.90 to 0.60] | -0.20 [-0.20 to 2.00]

71. Secondary Outcome: Bone Mineral Density (BMD), Total Body
Description: BMD as measured by dual-energy x-ray absorptiometry (DXA)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: grams per square centimeter
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
grams per square centimeter | 1.22 [1.18 to 1.27] | 1.22 [1.14 to 1.36]

72. Secondary Outcome: T-Score Femur Total Mean
Description: as for outcome 67
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
score on a scale | -0.10 [-0.93 to 0.02] | -0.80 [-1.25 to 0.50]

73. Secondary Outcome: T-Score Femur Total Mean
Description: as for outcome 67
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
score on a scale | -0.20 [-0.75 to 0.25] | -0.45 [-1.12 to 0.58]

74. Secondary Outcome: T-Score Femur Neck Mean
Description: as for outcome 67
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
score on a scale | -0.70 [-1.50 to 0.18] | -0.90 [-1.12 to -0.28]

75. Secondary Outcome: T-Score Femur Neck Mean
Description: as for outcome 67
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
score on a scale | -0.60 [-1.05 to 0.30] | -0.65 [-1.25 to -0.38]

76. Secondary Outcome: Bone Mineral Density (BMD), Femur Neck Mean
Description: BMD as measured by dual-energy x-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: grams per square centimeter
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
grams per square centimeter | 1.00 [0.94 to 1.11] | 0.99 [0.91 to 1.03]

77. Secondary Outcome: Bone Mineral Density (BMD), Femur Neck Mean
Description: BMD as measured by dual-energy x-ray absorptiometry (DXA)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: grams per square centimeter
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 12 | 9
grams per square centimeter | 0.98 [0.88 to 1.09] | 0.95 [0.92 to 1.04]

78. Secondary Outcome: Bone Mineral Density (BMD), Total Body
Description: BMD as measured by dual-energy x-ray absorptiometry (DXA)
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: grams per square centimeter
Arm/Group | Switch ART | Continue Current ART
Number analyzed (Participants) | 11 | 9
grams per square centimeter | 1.21 [1.14 to 1.27] | 1.21 [1.21 to 1.38]

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Switch ART | Continue Current ART
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT03348163/Prot_SAP_001.pdf